CLINICAL TRIAL: NCT00505973
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of SCA-136 Administered Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating the Safety and Tolerability of SCA-136 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3153A1-1114
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: SCA-136

SUMMARY:
This study is being conducted to assess the safety and tolerability of ascending multiple oral doses of SCA-136 administered to healthy Japanese male subjects.

ELIGIBILITY:
Inclusion criteria:

* Healty Japanese men willing to use a medically acceptable form of contraception.

Exclusion criteria:

* Any significant disease
* Positive urine drug screen
* Increased liver function tests
* Use of prescription drugs.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2007-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, safety laboratory results, vital signs, and ECGs will be used to monitor subject safety.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Ikebukuro, Toshima-ku, Japan